CLINICAL TRIAL: NCT05350917
Title: A Single-arm, Prospective, Open-label Clinical Study of Tislelizumab Combined With DisitamabVedotin and Pyrotinib Maleate in HER2-positive or Mutated Advanced Colorectal Cancer Who Failed Standard Therapy
Brief Title: Study of Tislelizumab Combined With DisitamabVedotin and Pyrotinib Maleate in HER2-positive or Mutated Advanced Colorectal Cancer Who Failed Standard Therapy
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The First Affiliated Hospital of Zhengzhou University (Other)
Collaborators: BeiGene (Industry); Jiangsu Hengrui Pharmaceutical Co., Ltd. (Industry); RemeGen Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Hong Zong, Department of Oncology, The First Affiliated Hospital of Zhengzhou University, The First Affiliated Hospital of Zhengzhou University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RCVDTYPEC024
Record Dates: First submitted 2022-02-17; First posted 2022-04-28 (Actual); Last update posted 2022-05-17 (Actual); Status verified 2022-05

CONDITIONS: HER2-positive or Mutated Advanced Colorectal Cancer
Keywords: HER2-positive or Mutated; Advanced Colorectal Cancer; failure of standard treatment; Tislelizumab Combined With DisitamabVedotin and Pyrotinib Maleate; PD-1 inhibitors+ADC+TKI
MeSH Terms: interventions — tislelizumab

STUDY DESIGN:
Intervention Model Description: A single-arm, prospective, open-label clinical study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tislelizumab Combined With DisitamabVedotin and Pyrotinib Maleate (Experimental): One arm study
  Interventions: Drug: Tislelizumab

INTERVENTIONS:
Drug: Tislelizumab — Tislelizumab: 200 mg, d1, intravenous infusion (ivgtt) administration, 21 days as a cycle.
  DisitamabVedotin : 2mg/kg, d1, intravenous drip (ivgtt) administration, 21 days as a cycle.
  Pyrotinib maleate tablets: 320 mg each time, Qd, orally administered within 30 minutes after breakfast, 21 days as a cycle.
  Continuous administration until disease progression, death, toxicity intolerance, withdrawal of informed consent, or other reasons specified in the protocol; for patients who still benefit after comprehensive evaluation after initial disease progression, the investigator may decide whether to continue the treatment with the experimental drug .
  Other Names: DisitamabVedotin; Pyrotinib maleate

SUMMARY:
This study will explore the efficacy and safety of tislelizumab (PD1 inhibitor) combined with DisitamabVedotin (ADC) and pyrotinib maleate (TKI) in the treatment of HER2-positive or mutated advanced colorectal cancer who have failed standard therapy .

ELIGIBILITY:
Inclusion Criteria：

* Colorectal cancer patients aged ≥18 years and ≤75 years old;
* ECOG score 0~1 points;
* Pathologically confirmed HER2 amplification-positive or mutated patients with advanced colorectal cancer who have failed or are intolerant of first-line therapy;
* Note: HER2 amplification positive means that in the pathological detection/recheck of the primary tumor or metastases conducted by the pathology department of our hospital, at least one tumor cell immunohistochemical staining intensity is 3+ or immunohistochemical staining intensity is 2+ and has been Fluorescence in situ hybridization [FISH] confirmed positive or NGS confirmed advanced colorectal cancer patients with HER2 gene amplification or mutation.
* According to RECIST1.1 criteria, there is at least one measurable target lesion, and tumor imaging evaluation is performed within 28 days before the first dose;
* Expected survival time ≥ 12 weeks;
* Major organ function is normal, that is, the following criteria are met:

  1. The blood routine examination standards must meet: ANC ≥1.5×109/L; PLT ≥90×109/L; Hb ≥90g/L (no blood transfusion within 14 days);
  2. Biochemical examinations should meet the following criteria: ALB≥30g/L; (no ALB transfusion within 14 days); TBIL≤Upper limit of normal (ULN); ALT and AST≤2.5 times upper limit of normal (ULN), if there is liver metastasis , then ALT and AST≤5ULN; alkaline phosphatase≤2.5 times the upper limit of normal (ULN); BUN and Cr≤1.5×ULN and creatinine clearance rate≥50 mL/min (CockcroftGault formula);
  3. Cardiac ultrasound and echocardiography: left ventricular ejection fraction (LVEF≥50%);(4) QT interval (QTcF) corrected by Fridericia method of 18-lead ECG in females <470 ms;
* For premenopausal or surgically sterilized female patients: consent to abstinence or use of effective contraception during treatment and for at least 7 months after the last dose of study treatment;
* Voluntarily join the study and sign the informed consent

Exclusion Criteria:

* Patients who have not received first-line standard therapy;
* Previous antitumor therapy or radiation therapy for any other malignant tumor;
* concurrently receiving anti-tumor therapy in other clinical trials, including endocrine therapy, bisphosphonate therapy, and immunotherapy;
* Has undergone major surgical procedures not related to colorectal cancer within 4 weeks prior to enrollment, or the patient has not fully recovered from such surgical procedures;
* Serious heart disease or discomfort, including but not limited to the following:

  * Diagnosed history of heart failure or systolic dysfunction (LVEF < 50%)
  * High-risk uncontrolled arrhythmias, such as atrial tachycardia, resting heart rate >100 bpm, significant ventricular arrhythmia (eg, ventricular tachycardia), or higher-grade AV block (ie, Mobitz II second-degree AV block or third-degree AV block)
  * Angina pectoris requiring antianginal drug treatment
  * Clinically significant heart valve disease
  * ECG showing transmural myocardial infarction
  * Poorly controlled hypertension (systolic blood pressure > 180 mmHg and/or diastolic blood pressure > 100 mmHg)
* Inability to swallow, bowel obstruction, or other factors that interfere with drug taking and absorption;
* Known history of allergy to the drug components of this regimen; history of immunodeficiency, including HIV positive test, or other acquired or congenital immunodeficiency diseases, or a history of organ transplantation;
* Pregnant or lactating female patients, female patients of childbearing potential with a positive baseline pregnancy test, or patients of childbearing age who are unwilling to take effective contraceptive measures throughout the trial period and within 7 months after the last study drug;
* have serious comorbidities or other comorbidities that would interfere with planned treatment, orAny other conditions for which the patient was deemed unsuitable for participation in this study by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-06-20 (Estimated); Primary Completion 2025-06-20 (Estimated); Study Completion 2026-06-20 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | Up to 24 months
  It is defined as the number of subjects with the best response effect as complete remission (CR) or partial remission (PR) during the period from the start of the subjects receiving the treatment regimen of this study to the progression of the subjects' disease in the total number of subjects in the analysis data set. percentage of the population（%）.

SECONDARY OUTCOMES:
Disease Control Rate (DCR) | Up to 24 months
  Defined as the number of subjects whose tumors shrank or remained stable for a certain period of time from receiving the treatment regimen of this study to the progression of the subject's disease, including complete remission (CR) and partial remission (PR) in the analysis data set percentage of the total population（%）.
Progression Free Survival (PFS) | Up to 24 months
  Defined as the time from randomization to tumor progression in any aspect or death from any cause（Unit: month）.
  Assessed according to RECIST 1.1 criteria, analysis of this indicator included tumor evaluation results during study treatment and follow-up. If the patient has several indicators that can be judged as PD, the first indicator will be used for PFS analysis; recurrence, new lesions or death are considered to have reached the end of the study, and the patient is treated with other systemic or target-targeted anti-PD. Tumor treatment is also considered tumor progression.
Overall survival (OS) | Up to 24 months
  Defined as the time from randomization to death from any cause（Unit: month）.
Drug-Related Safety Indicators | Up to 24 months
  Exposure to the investigational drug and incidence, nature, and severity of adverse events, including serious adverse events（n，%）。
Study on the mechanism of drug resistance after progression | Up to 24 months
  Changes in HER2 status, HER2 gene, and HER2-related signaling pathways before and after treatment.
  Note: HER2 positive means that in the pathological detection/recheck of the primary or metastatic lesions performed by the pathology department, at least one tumor cell immunohistochemical staining intensity of 3+ or immunohistochemical staining intensity of 2+ and fluorescence in situ hybridization Technical [FISH] confirmed positive or NGS confirmed advanced colorectal cancer patients with HER2 gene amplification or mutation.

IPD SHARING:
Plan to Share IPD: No